CLINICAL TRIAL: NCT01241084
Title: Beneficial Effects of Lactobacillus Reuteri DSM 17938 Supplementation on the Airways Allergic Inflammation of Asthmatic Children
Brief Title: Beneficial Effects of Lactobacillus Reuteri DSM 17938 Supplementation on Asthmatic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Prof. Michele Miraglia del Giudice, MD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Lr_Asthma
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Airways Allergic Inflammation of Asthmatic Children
Keywords: asthmatic children
MeSH Terms: interventions — Leukotriene Antagonists

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Antileukotrienes+Placebo
  Interventions: Dietary Supplement: Antileukotrienes + Placebo
- Lactobacillus reuteri (Active Comparator): Antileukotrienes+Lactobacillus reuteri
  Interventions: Dietary Supplement: Antileukotrienes + Lactobacillus reuteri

INTERVENTIONS:
Dietary Supplement: Antileukotrienes + Lactobacillus reuteri — Montelukast (5mg/die) + 1000000000 CFU per day (5 drops) for 2 months
  Arms: Lactobacillus reuteri
Dietary Supplement: Antileukotrienes + Placebo — Montelukast (5mg/die) + 5 drops of placebo daily for 2 months
  Arms: Placebo

SUMMARY:
Objective The aim of the trial is to evaluate the beneficial effects of the oral administration of the probiotic L. Reuteri (Reuterin®) on the airways allergic inflammation in children with mild to moderate persistent asthma.

Study design This is a randomized, double-blind, placebo controller trial. 50 children will be enrolled (age range 6-14 years), affected by mild to moderate persistent asthma based on the GINA Guidelines and allergic to acarus (Dermatophagoides farinae and D. pteronyssinus ++/+++). At the enrollment period all children have to show asthmatic symptoms and to be under antileukotrienes treatment (Montelukast 5mg/die) based on the GINA Guidelines. Any inhaling corticosteroids therapies have to be stopped 8 weeks before the trial beginning.

Patients will be randomly divided into 2 treatment groups:

Group A: 25 patients will take antileukotrienes + L. reuteri drops (108 CFU = 5 drops daily).

Group B: 25 patients will take antileukotrienes + placebo. At the enrollment period (T0), after the 1st and the 2nd month of supplementation (T1 and T2), and also 1 month after the supplementation end (T3), all patients will be clinically evaluated through spirometry, FeNO determination and exhale condensate analysis.

During the entire trial period the number of asthmatic exacerbations and the use of beta-2 antagonists will be monitored by a diary properly examined at T1, T2 and T3.

All children will be enrolled at the Asthma and Infant Respiratory Physiopathology unit "Michele Miraglia del Giudice" of the "F. Fede" Pediatric Department.

The analysis of the inflammatory markers on the exhaled condensate will be performer at T1, T2 and T3 in the Pharmacology unit of the Experimental Medicine Department.

During the trial it will be possible to administer only salbutamole MDI if it needed. If patients will be administered with any systemic corticosteroids they will exit from the trial.

At the enrolment period all patients will receive the completed information on the trial and the informed consent will be properly signed.

ELIGIBILITY:
Inclusion Criteria:

* Children with age range 6-14 years
* Informed consent signed

Exclusion Criteria:

* Participation to other clinical trials
* Informed consent not signed

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Beneficial effects of Lactobacillus reuteri supplementation on asthmatic children | two months
  At the enrollment period all children have to show asthmatic symptoms and to be under antileukotrienes treatment (Montelukast 5mg/die) based on the GINA Guidelines. .
  At the enrolment period (T0), after the 1st and the 2nd month of supplementation (T1 and T2), and also 1 month after the supplementation end (T3), all patients will be clinically evaluated through spirometry, FeNO determination and exhale condensate analysis.
  During the entire trial period the number of asthmatic exacerbations and the use of beta-2 antagonists will be monitored by a diary properly examined at T1, T2 and T3.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Miraglia del Giudice, MD, Principal Investigator — AOU "Federico II" di Napoli
Locations (1):
- AOU "Federico II" di Napoli, Napoli, Italy